CLINICAL TRIAL: NCT04265235
Title: EXerCise Intervention in cholesTatic LivEr Disease: The EXCITED Study
Acronym: EXCITED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID pandemic. Recruited 31 out of target 40 patients.
Sponsor: University of Birmingham (Other)
Collaborators: University Hospital Birmingham NHS Foundation Trust (Other); Intercept Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Matthew Armstrong, Consultant in Liver and Transplant Medicine, Honorary Clinical research Fellow and Principal Investigator, University of Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RRK6589
Record Dates: First submitted 2020-02-06; First posted 2020-02-11 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Primary Biliary Cholangitis
Keywords: Exercise; Fatigue; Liver
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Motor Activity; Fatigue

STUDY DESIGN:
Intervention Model Description: Single-arm Exercise Intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-based Exercise Program (Experimental): 12-weeks, remotely monitored home-based exercise program consisting or aerobic and resistance exercise
  Interventions: Other: Home-based exercise program

INTERVENTIONS:
Other: Home-based exercise program — see 'arm' section

SUMMARY:
A prospective, single centre, single-arm, pilot study investigating the safety and efficacy of a 12-week remotely-monitored home-based exercise program in patients with refractory fatigue (based on PBC-40 Quality of Life measure) secondary to Primary Biliary Cirrhosis.

DETAILED DESCRIPTION:
Recruitment from the research nurse-led PBC clinic: Eligibility screen followed by recruitment letters being sent to patients.

The outpatient clinic review by the liver specialist physiotherapist (week 0):

Patients will undergo a baseline assessment of quality of life, anthropometry, functional capacity (with validated tools including the incremental shuttle walk test and short performance battery test) and exercise tolerance. At the same visit, patients will be prescribed and trained to perform the individualised Home-based Exercise Program. Patients will be provided with an accelerometer to assess daily step count and a symptoms/side effects diary.

Six weeks of telephone support (weeks 0-6):

Patients will be telephoned weekly over a period of 6 weeks, in order to evaluate compliance with therapy and any difficulties encountered. At each phone call, the daily step count and the intensity of the resistance-exercises will be adjusted to the patients ability.

The outpatient clinic review by the liver specialist physiotherapist (week 6 +/- 5 days): Reassessment of baseline parameters of quality of life, functionality and exercise tolerance; and modification of step count targets and resistance-exercise intervention as needed.

The outpatient clinic review by the liver specialist physiotherapist (week 12 +/- 5 days): Reassessment of baseline parameters of quality of life, functionality and exercise tolerance; and modification of step count targets and resistance-exercise intervention as needed.

Validate the efficacy of exercise intervention: Given that the goal is to improve fatigue-related symptoms and thus patient quality of life, the investigators will determine the interim efficacy and longevity of intervention using a multi-modal patient-reported outcome approach. This will principally be through changes in validated quality of life (QoL) scoring measures at baseline and during sequential study visits; including the fatigue domain of the PBC-40 QoL measure (primary outcome measure), in addition to the relevant PBC-40 domains of cognitive, social, emotional and overall symptom burden; the Hospital Anxiety and Depression Scale (HADS); Epworth Sleepiness Scale to assess daytime somnolence; Patient-Reported Outcomes Measurement Information System Health Assessment Questionnaire (PROMIS-HAQ®) to assess functional status, and the Cognitive Failure questionnaire (COGFAIL) to determine cognitive functionality.

All data will be collated onto a standardised clinical case record form. Outcomes will be audited after 6 months to determine whether the intervention has proven beneficial to patients, and whether improvements in functional status correlate with changes in fatigue and QoL scores

ELIGIBILITY:
Inclusion Criteria:

* 18 Years Old
* A confirmed diagnosis of PBC through clinical observation as per guidance of BSG/ EASL
* Fatigue Impact Scale >40
* Access to a SMART Phone or Computer

Exclusion Criteria:

* Decompensated PBC with the following clinical signs:
* Moderate Ascites
* A Bilirubin of >50
* Variceal Bleed < 6 Months
* Encephalopathic
* Refractory Pruritis (Judged by PI)
* Cardiovascular Instability (Judged by PI)
* Untreated Vitamin Deficiency
* Untreated hypothyroidism
* Untreated Coeliac Disease
* WHO Performance Status > 3
* History of Unexplained Falls

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-04-07 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Change in PBC-40 Quality of Life for Primary Biliary Cirrhosis | 12 weeks
  PBC-40 is a quality of life questionnaire (validated) with the domains of cognitive, social, emotional and overall symptom burden. 40 questions, each scored on a scale of 1 to 5 (where 1 = least impact, 5 = greatest impact)

SECONDARY OUTCOMES:
Health Anxiety Depression Score (HADS) | 12 weeks
  Questionnaire - out of 24. higher score means worse depression and anxiety
hand grips strength (kg) | 12 weeks
  measures of muscle strength
liver frailty index | 12 weeks
  index based on hand grip strength, chair stands, balance. higher the value the more frail.

CONTACTS AND LOCATIONS:
Locations (1):
- Liver Unit, University Hospital Birminghmam, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Freer A, Williams FR, Durman S, Hayden J, Armstrong MJ, Trivedi PJ. A home-based exercise programme attenuates fatigue in primary biliary cholangitis: Results from the EXCITED clinical trial. JHEP Rep. 2024 Sep 6;6(12):101210. doi: 10.1016/j.jhepr.2024.101210. eCollection 2024 Dec. PMID 39640219
- [Derived] Freer A, Williams F, Durman S, Hayden J, Trivedi PJ, Armstrong MJ. Home-based exercise in patients with refractory fatigue associated with primary biliary cholangitis: a protocol for the EXerCise Intervention in cholesTatic LivEr Disease (EXCITED) feasibility trial. BMJ Open Gastroenterol. 2021 Mar;8(1):e000579. doi: 10.1136/bmjgast-2020-000579. PMID 33707216